CLINICAL TRIAL: NCT07138417
Title: Investigating the Therapeutic Mechanism of Compassion-Based Family Intervention for Adolescents With Emotional Disorders and Their Parents
Brief Title: The Therapeutic Mechanism of Compassion-Based Family Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing HuiLongGuan Hospital (Other)
Responsible Party: Principal Investigator, Xiang Yang Zhang, Professor, Beijing HuiLongGuan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CASPsy8
Record Dates: First submitted 2025-07-30; First posted 2025-08-22 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Emotional Disorder
Keywords: Emotional disorder; adolescents; compassion; parents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compassion-based family intervention group (Experimental): A six-week compassion-based family intervention will be conducted , consisting of one session per week. Each 120-minute session included the following components: Introduction (10 min); Cognitive Intervention (50 min); Group Activities & Parent-Child Interaction (50 min); Summary (10 min).
  Additionally, during the six-week intervention period, families will complete supplementary exercises, including three relaxation meditation sessions per week and three emotional journal per week.
  Interventions: Other: Compassion-Based Family Therapy
- Waiting list control group (No Intervention): The waiting list control group waited for 6 weeks after the baseline measurement for the post-test, and then conducted the same intervention.

INTERVENTIONS:
Other: Compassion-Based Family Therapy — Draw ideas from traditional Chinese culture, the investigators have developed the compassion-based family intervention therapy to improve the mental health of both parents and children by enhancing their synchronization.
  The 6-week program followed a progressive thematic structure. Week 1 focuses on introduction and connection, themed "Setting Sail: The Additions and Subtractions for a Happy Family." Weeks 2 and 3 address self-compassion: Week 2 is themed "Self-compassion: Embrace yourself with compassion here and now."; Week 3 is themed "Self-compassion: Accepting "growing pains."." Weeks 4 and 5 explored developing compassion for others: Week 4 is themed "Listening to the heart: Enhancing communication, bringing us closer."; Week 5 is themed "Building a harbor together: Managing conflict, creating happiness" Week 6 involves integration and review, themed "Integrating knowledge and action: Practicing compassion, lighting the path forward."
  Arms: Compassion-based family intervention group

SUMMARY:
1. To investigate the correlations between self-compassion-related variables in parents of adolescents with emotional disorders and parenting stress as well as self-stigmatization; and the correlations between self-compassion-related variables and the severity of depressive and anxiety symptoms in adolescents.
2. To evaluate the effectiveness of a Compassion-Focused Family Intervention in increasing self-compassion among adolescents and their parents, and in reducing parenting stress, self-stigmatization, and the severity of adolescent depression and anxiety.
3. To explore the neural and physiological mechanisms underlying the therapeutic effects of the compassion intervention on parent-child interactions, using functional near-infrared spectroscopy (fNIRS) hyperscanning and wearable wristband devices.

DETAILED DESCRIPTION:
This study plans to recruit 120 families (each consisting of a 12-18-year-old adolescent with emotional disorders and their parents), and randomly divide them into an intervention group and a control group, with 60 pairs in each group. The intervention group received a 6-week compassion-based family intervention, once a week for 120 minutes each time, accompanied by family exercises including meditation training and emotional journal. The waiting list control group waited for 6 weeks after the baseline measurement for the post-test, and then conducted the same intervention.

The study adopted multi-dimensional assessment: at five time points including baseline, immediately after the intervention, and 3, 6 month follow-up, the psychological state of parents and children was measured through psychological scales (such as the Children's Depression Inventory Scale and the Child-Parent Relationship Scale). At the same time, near-infrared hyperscanning technology was used to record the synchronization of brain signals when parents and children watched emotional videos (2 positive/neutral/negative segments each) (analyzing neural synchronization in the 0.02-0.10Hz frequency band), and a wearable bracelet was used to monitor physiological indicators such as heart rate variability. Data analysis will examine the effect of intervention on enhancing parents' self-compassion level, reducing parenting pressure and symptoms of depression and anxiety in adolescents, and explore the association mechanism between parent-child neural synchrony changes and intervention effects. Ultimately, it will verify the effectiveness of compassion therapy in improving the mental health of families of adolescents with emotional disorders.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12-18 years
* Required scores at enrollment: 17-item Hamilton Depression Rating Scale (HAMD-17) total score≥17 and ≤30; or Hamilton Anxiety Rating Scale (HAMA) total score ≥18 and ≤29
* Required scores at enrollment: The item 3 score of HAMD-17 (suicide) ≤2
* No clear suicide plan or recent suicide attempt history; with consistent feedback from parents/guardians
* No history of severe psychotic symptoms or manic episodes
* No history of substance abuse
* Parent(s) willing to participate
* Absence of psychotic symptoms, no contraindications for MRI, and no major physical illnesses, etc.

Exclusion Criteria:

* Adolescents diagnosed with a major psychiatric disorder (e.g., schizophrenia)
* Adolescents presenting with comorbid psychotic features
* Adolescents assessed as having suicide risk
* Parents who are illiterate (lacking reading and writing ability)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Perceived emotional synchrony | baseline, immediately after the intervention, and 3, 6 month follow-up
  Using the score of Perceived Emotional Synchrony Scale to assess perceived emotional synchrony of parents and children respectively.
  Perceived emotional synchrony scale (16-item version): items rated 1-7; the investigators report mean subscale scores (range 1-7) for Emotional Communion (items 1, 4, 5, 7, 8, 11, 14, 15) and Felt Unity (items 2, 3, 6, 9, 10, 12, 13, 16). Higher scores indicate greater perceived emotional synchrony (better outcome).
Self-Compassion | baseline, immediately after the intervention, and 3, 6 month follow-up
  Using the Self-Compassion Scale to assess self-compassion levels of parents and children respectively.
  Self-Compassion Scale (SCS): 26 items rated 1-5; the investigators report the mean score (range 1-5). Higher scores indicate greater self-compassion (better outcome).
Fears of Compassion | baseline, immediately after the intervention, and 3, 6 month follow-up
  Using the Fears of Compassion Scales to assess fears of compassion levels of parents and children respectively.
  Fears of Compassion Scales (FCS): three subscales rated 0-4 - Fear of Compassion for Self (15 items; total 0-60), Fear of Compassion for Others (10 items; total 0-40), and Fear of Receiving Compassion from Others (13 items; total 0-52). Higher scores indicate greater fear of compassion (worse outcome).
Parenting Stress | baseline, immediately after the intervention, and 3, 6 month follow-up
  Using the Parenting Stress Index-Short Form to assess parenting stress. Parenting Stress Index-Short Form (PSI-SF): 36 items rated 1-5; the investigators report the total score (range 36-180). Higher scores indicate greater parenting stress (worse outcome).
Children's depression levels | baseline, immediately after the intervention, and 3, 6 month follow-up
  Using the Children's Depression Inventory scale to assess children's depression levels.
  Children's Depression Inventory (CDI): 27 items rated 0-2; the investigators report the total score (range 0-54). Higher scores indicate more severe depressive symptoms (worse outcome).
Children's anxiety levels | baseline, immediately after the intervention, and 3, 6 month follow-up
  Using the Beck Anxiety Inventory to assess children's anxiety levels. Beck Anxiety Inventory (BAI): 21 items rated 0-3; the investigators report the total score (range 0-63). Higher scores indicate more severe anxiety (worse outcome).
Oxy-hemoglobin concentration change (ΔHbO) | baseline, immediately after the intervention, and 3, 6 month follow-up
  Functional near-infrared spectroscopy (fNIRS) hyperscanning was employed to measure wavelet transform coherence (WTC) between parents and children during an emotional video task. The primary signals of interest were the concentration changes of oxy-hemoglobin (ΔHbO) and deoxy-hemoglobin (ΔHbR). ΔHbO and ΔHbR signals were preprocessed before WTC analysis. The WTC frequency band was set at 0.02-0.10 Hz to assess brain signal synchrony in time-frequency domains, providing higher sensitivity than traditional correlation coefficients. Higher coherence values indicated stronger neural synchrony.
Deoxy-hemoglobin concentration change (ΔHbR) | baseline, immediately after the intervention, and 3, 6 month follow-up
  Functional near-infrared spectroscopy (fNIRS) hyperscanning was employed to measure wavelet transform coherence (WTC) between parents and children during an emotional video task. The primary signals of interest were the concentration changes of oxy-hemoglobin (ΔHbO) and deoxy-hemoglobin (ΔHbR). ΔHbO and ΔHbR signals were preprocessed before WTC analysis. The WTC frequency band was set at 0.02-0.10 Hz to assess brain signal synchrony in time-frequency domains, providing higher sensitivity than traditional correlation coefficients. Higher coherence values indicated stronger neural synchrony.
Heart rate variability (HRV) | baseline, immediately after the intervention, and 3, 6 month follow-up
  Heart rate variability (HRV) metrics in parents and children were measured using wearable wristbands (Huawei Band 8) throughout both the emotional video task and group intervention sessions.

SECONDARY OUTCOMES:
Parenting styles | baseline, immediately after the intervention, and 3, 6 month follow-up
  Using the Parenting Scale-7 to assess parenting styles. Parenting Scale-7 (PS-7): 7 items rated 1-7; the investigators report the mean score (range 1-7). Higher scores indicate more dysfunctional parenting practices (worse outcome).
Parenting styles in children's view | baseline, immediately after the intervention, and 3, 6 month follow-up
  Using the Egna Minnen av Barndoms Uppfostran to assess the parenting styles in children's view.
  Egna Minnen av Barndoms Uppfostran (EMBU; "My Memories of Upbringing"), 21-item version: items rated 1-4; the investigators report summed subscale scores for Rejection (items 1, 4, 7, 12, 14, 19), Emotional Warmth (items 2, 6, 9, 11, 13, 17, 21), and Overprotection (items 3, 5, 8, 10, 15R, 16, 18, 20), with item 15 reverse-scored. Higher Rejection and Overprotection indicate worse outcomes, whereas higher Emotional Warmth indicates better outcomes.
Parent-child relationships in parents' view | baseline, immediately after the intervention, and 3, 6 month follow-up
  Using the Child-Parent Relationship Scale, 10-item scale to assess the Parent-child relationships from the perspective of parents.
  Child-Parent Relationship Scale, 30-item version (CPRS): items rated 1-5; the investigators report mean subscale scores (range 1-5) for Closeness, Conflict, and Dependence. Higher Closeness indicates a better relationship (better outcome), whereas higher Conflict and higher Dependence indicate worse outcomes.
Parent-child relationships in children's view | baseline, immediately after the intervention, and 3, 6 month follow-up
  Using the Remembered Relationship with Parents, 10-item scale to assess the Parent-child relationships from the perspective of children.
  Remembered Relationship with Parents, 10-item scale (RRP10): 10 items rated 0-4; the investigators report the total score (range 0-40). Higher scores indicate more negative remembered relationships with parents (worse outcome).
Nonclinging to Ego | baseline, immediately after the intervention, and 3, 6 month follow-up
  Using the Nonclinging to Ego Scale to assess nonclinging to ego levels of parents and children respectively.
  Nonclinging to Ego Scale (NES): 33 items rated 1-6; the investigators report the total score (range 33-198). Higher scores indicate greater nonattachment to self (better outcome).
Parental self-stigmatization | baseline, immediately after the intervention, and 1, 3, 6 month follow-up
  Using the Self-Stigma in Relatives of people with Mental Illness Scale to assess the parental self-stigmatization.
  Self-Stigma in Relatives of people with Mental Illness Scale (SSRMI): 30 items rated 1-5; the investigators report the mean score (range 1-5). Higher scores indicate greater self-stigma among relatives (worse outcome).
Perceived Criticism | baseline, immediately after the intervention, and 3, 6 month follow-up
  Using the Perceived Criticism Measure to assess the parent' perceived criticism levels.
  Perceived Criticism Measure (PCM): items rated 1-10; the investigators report the mean score (range 1-10). Higher scores indicate greater perceived criticism (worse outcome).
Family Expressiveness | baseline, immediately after the intervention, and 3, 6 month follow-up
  Using the Family Expressiveness Questionnaire to assess the family expressiveness.
  Family Expressiveness Questionnaire (FEQ): 20 items rated 1-9; the investigators report the mean score (range 1-9). Higher scores indicate more frequent family emotional expressiveness; when reporting Positive vs. Negative Expressiveness subscales, higher Positive is considered better and higher Negative is considered worse.
Emotion Regulation | baseline, immediately after the intervention, and 3, 6 month follow-up
  Using the Emotion Regulation Questionnaire, 6-item version to assess the emotion regulation levels of parents and children respectively.
  Emotion Regulation Questionnaire, 6-item version (ERQ-6): items rated 1-7; the investigators report mean subscale scores (range 1-7) for Cognitive Reappraisal (4 items) and Expressive Suppression (2 items). Higher Reappraisal indicates more frequent use of cognitive reappraisal (typically better outcome), whereas higher Suppression indicates more frequent use of expressive suppression (typically worse outcome).
Concise Chinese Level of Expressed Emotion | baseline, immediately after the intervention, and 3, 6 month follow-up
  Using the Concise Chinese Level of Expressed Emotion Scale to assess the concise Chinese level of expressed emotion of children.
  Concise Chinese Level of Expressed Emotion Scale (CCLEES): 12 items rated 1-4; the investigators report the mean score (range 1-4). Higher scores indicate higher expressed emotion (typically associated with worse outcomes).
Parental Burnout | baseline, immediately after the intervention, and 3, 6 month follow-up
  Using the Parental Burnout Assessment to assess the parental burnout level. Parental Burnout Assessment (PBA): 23 items rated 0-6; the investigators report the total score (range 0-138). Higher scores indicate greater parental burnout (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Wang, Ph.D, Principal Investigator — Institute of Psychology, Chinese Academy of Science
Locations (2):
- China (2):
  - Anhui Mental Health Center, Hefei, Anhui
  - Institute of Psychology, Chinese Academy of Sciences, Beijing, Beijing

IPD SHARING:
Plan to Share IPD: No
Data with be available on request